CLINICAL TRIAL: NCT02635828
Title: Studying the Effectiveness of Triple Therapy With Palonosetron, Dexamethasone and Promethazine for Prevention of Post Operative Nausea and Vomiting in High Risk Patients Undergoing Neurological Surgery and General Anesthesia
Brief Title: Effectiveness of Triple Therapy With Palonosetron for PON Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Sergio Bergese, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008H0170
Record Dates: First submitted 2015-12-08; First posted 2015-12-21 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Palonosetron; Craniotomy; Nausea; Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Palonosetron; Dexamethasone; Calcium Dobesilate; Promethazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple therapy PONV prophylaxis (Experimental): At induction of anesthesia, a triple therapy of palonosetron 0.075 mg IV, dexamethasone 10 mg IV and promethazine 25 mg IV was given as PONV prophylaxis.
  Interventions: Drug: Palonosetron 0.075 mg IV; Drug: Dexamethasone 10 mg IV; Drug: Promethazine 25 mg IV

INTERVENTIONS:
Drug: Palonosetron 0.075 mg IV — At induction of anesthesia, palonosetron 0.075 mg IV was given as PONV prophylaxis.
  Other Names: Aloxi
Drug: Dexamethasone 10 mg IV — At induction of anesthesia, dexamethasone 10 mg IV was given as PONV prophylaxis.
  Other Names: Decadron
Drug: Promethazine 25 mg IV — At induction of anesthesia, promethazine 25 mg was given as PONV prophylaxis.
  Other Names: Phenergan

SUMMARY:
Postoperative nausea and vomiting (PONV) is a displeasing experience that distresses surgical patients during the first 24 hours after a surgical procedure. The incidence of postoperative nausea occurs in about 50%, the incidence of postoperative vomiting is about 30%, and in high-risk patients, the PONV rate could be as high as 80%. Therefore, the study design of this single arm, non-randomized, pilot study assessed the efficacy and safety profile of a triple therapy combination with palonosetron, dexamethasone and promethazine to prevent PONV in patients undergoing craniotomies under general anesthesia.

DETAILED DESCRIPTION:
At induction of anesthesia, a triple therapy of palonosetron 0.075 mg IV, dexamethasone 10 mg IV and promethazine 25 mg IV was given as PONV prophylaxis. After surgery, subjects were transferred to the surgical intensive care unit (SICU) or post anesthesia care unit as clinically indicated. Ondansetron 4 mg IV was administered as primary rescue medication to subjects with PONV symptoms. PONV was assessed and collected every 24 hours for 5 days via direct interview and/or medical charts review.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 85 years of age, of any race or gender. With an American Society of Anesthesiologist (ASA) physical status of I to III who are scheduled to undergo neurological surgery requiring opening of the cranium and Dura matter under general anesthesia, at Ohio State University Medical Center and who consent in writing to participating in this study.
* Post operative hospitalization expected to last at least 72 hours.
* Subjects whose surgery is expected to require at least 1 hours of general anesthesia
* Subjects who have a negative serum or urine pregnancy test within 1 day of surgery or who have been surgically sterilized or are postmenopausal.

Exclusion Criteria:

* Subjects who are prisoners, pregnant, mentally ill, under the age of 18 or over the age of 85, ASA classification of V, alcohol or drug abusers.
* Subjects with known hypersensitivity to any 5-HT3 antagonist, to any agent that is part of the anesthesia regimen, or to other medications to be administered under this protocol.
* Subjects who are breastfeeding.
* Subjects who have had retching/vomiting or moderate to severe nausea in the 24 hours prior to anesthesia or suffer chronic nausea and/or vomiting
* Subjects who have been treated with any drug or other treatment with anti-emetic efficacy within the last 24 hours prior to the start of treatment.
* Subjects who have participated in a clinical trial of an investigational drug within 30 days prior to surgery.
* Subjects who are participating in any other clinical study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto A Uribe, M.D., Study Chair — Ohio State University

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Result] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Result] Kovac AL. Prevention and treatment of postoperative nausea and vomiting. Drugs. 2000 Feb;59(2):213-43. doi: 10.2165/00003495-200059020-00005. PMID 10730546
- [Result] Fabling JM, Gan TJ, El-Moalem HE, Warner DS, Borel CO. A randomized, double-blinded comparison of ondansetron, droperidol, and placebo for prevention of postoperative nausea and vomiting after supratentorial craniotomy. Anesth Analg. 2000 Aug;91(2):358-61. doi: 10.1097/00000539-200008000-00023. PMID 10910848
- [Result] Gan TJ, Meyer T, Apfel CC, Chung F, Davis PJ, Eubanks S, Kovac A, Philip BK, Sessler DI, Temo J, Tramer MR, Watcha M; Department of Anesthesiology, Duke University Medical Center. Consensus guidelines for managing postoperative nausea and vomiting. Anesth Analg. 2003 Jul;97(1):62-71, table of contents. doi: 10.1213/01.ane.0000068580.00245.95. PMID 12818945
- [Result] Audibert G, Vial V. [Postoperative nausea and vomiting after neurosurgery (infratentorial and supratentorial surgery)]. Ann Fr Anesth Reanim. 2004 Apr;23(4):422-7. doi: 10.1016/j.annfar.2004.01.005. French. PMID 15120791
- [Result] Manninen PH, Raman SK, Boyle K, el-Beheiry H. Early postoperative complications following neurosurgical procedures. Can J Anaesth. 1999 Jan;46(1):7-14. doi: 10.1007/BF03012507. PMID 10078396
- [Result] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Result] Sanger GJ, Andrews PL. Treatment of nausea and vomiting: gaps in our knowledge. Auton Neurosci. 2006 Oct 30;129(1-2):3-16. doi: 10.1016/j.autneu.2006.07.009. Epub 2006 Aug 24. PMID 16934536
- [Result] Habib AS, Gan TJ. Combination therapy for postoperative nausea and vomiting - a more effective prophylaxis? Ambul Surg. 2001 Jul;9(2):59-71. doi: 10.1016/s0966-6532(01)00103-2. PMID 11454483
- [Result] Ku CM, Ong BC. Postoperative nausea and vomiting: a review of current literature. Singapore Med J. 2003 Jul;44(7):366-74. PMID 14620731
- [Result] Habib AS, El-Moalem HE, Gan TJ. The efficacy of the 5-HT3 receptor antagonists combined with droperidol for PONV prophylaxis is similar to their combination with dexamethasone. A meta-analysis of randomized controlled trials. Can J Anaesth. 2004 Apr;51(4):311-9. doi: 10.1007/BF03018234. PMID 15064259
- [Result] Khalil S, Philbrook L, Rabb M, Wells L, Aves T, Villanueva G, Amhan M, Chuang AZ, Lemak NA. Ondansetron/promethazine combination or promethazine alone reduces nausea and vomiting after middle ear surgery. J Clin Anesth. 1999 Nov;11(7):596-600. doi: 10.1016/s0952-8180(99)00103-8. PMID 10624646
- [Result] Board T, Board R. The role of 5-HT3 receptor antagonists in preventing postoperative nausea and vomiting. AORN J. 2006 Jan;83(1):209-16, 219-20. doi: 10.1016/s0001-2092(06)60241-x. PMID 16528908
- [Result] Siddiqui MA, Scott LJ. Palonosetron. Drugs. 2004;64(10):1125-32; discussion 1133-4. doi: 10.2165/00003495-200464100-00006. PMID 15139789
- [Result] Rojas C, Stathis M, Thomas AG, Massuda EB, Alt J, Zhang J, Rubenstein E, Sebastiani S, Cantoreggi S, Snyder SH, Slusher B. Palonosetron exhibits unique molecular interactions with the 5-HT3 receptor. Anesth Analg. 2008 Aug;107(2):469-78. doi: 10.1213/ane.0b013e318172fa74. PMID 18633025
- [Result] Gralla R, Lichinitser M, Van Der Vegt S, Sleeboom H, Mezger J, Peschel C, Tonini G, Labianca R, Macciocchi A, Aapro M. Palonosetron improves prevention of chemotherapy-induced nausea and vomiting following moderately emetogenic chemotherapy: results of a double-blind randomized phase III trial comparing single doses of palonosetron with ondansetron. Ann Oncol. 2003 Oct;14(10):1570-7. doi: 10.1093/annonc/mdg417. PMID 14504060
- [Result] Aapro MS, Grunberg SM, Manikhas GM, Olivares G, Suarez T, Tjulandin SA, Bertoli LF, Yunus F, Morrica B, Lordick F, Macciocchi A. A phase III, double-blind, randomized trial of palonosetron compared with ondansetron in preventing chemotherapy-induced nausea and vomiting following highly emetogenic chemotherapy. Ann Oncol. 2006 Sep;17(9):1441-9. doi: 10.1093/annonc/mdl137. Epub 2006 Jun 9. PMID 16766588
- [Result] Candiotti KA, Kovac AL, Melson TI, Clerici G, Joo Gan T; Palonosetron 04-06 Study Group. A randomized, double-blind study to evaluate the efficacy and safety of three different doses of palonosetron versus placebo for preventing postoperative nausea and vomiting. Anesth Analg. 2008 Aug;107(2):445-51. doi: 10.1213/ane.0b013e31817b5ebb. PMID 18633022
- [Result] Kovac AL, Eberhart L, Kotarski J, Clerici G, Apfel C; Palonosetron 04-07 Study Group. A randomized, double-blind study to evaluate the efficacy and safety of three different doses of palonosetron versus placebo in preventing postoperative nausea and vomiting over a 72-hour period. Anesth Analg. 2008 Aug;107(2):439-44. doi: 10.1213/ane.0b013e31817abcd3. PMID 18633021
- [Derived] Bergese SD, Puente EG, Antor MA, Capo G, Yildiz VO, Uribe AA. The Effect of a Combination Treatment Using Palonosetron, Promethazine, and Dexamethasone on the Prophylaxis of Postoperative Nausea and Vomiting and QTc Interval Duration in Patients Undergoing Craniotomy under General Anesthesia: A Pilot Study. Front Med (Lausanne). 2016 Feb 2;3:1. doi: 10.3389/fmed.2016.00001. eCollection 2016. PMID 26870733

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 54 participants provided written consent for the study, and only 40 participants were randomized.
Groups:
- Triple Therapy PONV Prohylaxis: At induction of anesthesia, a triple therapy of palonosetron 0.075 mg IV, dexamethasone 10 mg IV and promethazine 25 mg IV was given as PONV prophylaxis.
  Palonosetron 0.075 mg IV: At induction of anesthesia, palonosetron 0.075 mg IV was given as PONV prophylaxis.
  Dexamethasone 10 mg IV: At induction of anesthesia, dexamethasone 10 mg IV was given as PONV prophylaxis.
  Promethazine 25 mg IV: At induction of anesthesia, promethazine 25 mg was given as PONV prophylaxis.
Period: Overall Study
Arm/Group | Triple Therapy PONV Prohylaxis
Started | 54
Completed | 40
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Triple Therapy PONV Prohylaxis
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: PONV Incidence
Description: The incidence of PONV
Time Frame: 24 hours after end of surgery
Population: Incidence of PONV
Measure: Number; unit: participants
Arm/Group | Triple Therapy PONV Prohylaxis
Number analyzed (Participants) | 40
participants | 12

2. Secondary Outcome: Incidence of Subjects Significant QTc Changes in the EKG
Description: The incidence of significant QTc prolongation was measured by comparing baseline EKG, 24 hours and 120 hours after surgery
Time Frame: 24 and 120 hours/discharge after end of surgery
Measure: Number; unit: participants
Arm/Group | Triple Therapy PONV Prohylaxis
Number analyzed (Participants) | 40
participants | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Triple Therapy PONV Prohylaxis
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Our study also presented certain limitations that should be mentioned. To begin with, the study was designed without a control group; therefore, we were not able to compare the results from this regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No